CLINICAL TRIAL: NCT04545593
Title: Building Community Capacity for Disability Prevention for Minority Elders - Renewal
Brief Title: Positive Minds Strong Bodies Implementation
Acronym: PMSB-E
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019P001292
Record Dates: First submitted 2020-09-04; First posted 2020-09-11 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Depression; Anxiety; Physical Disability
Keywords: Minority Elders
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research staff conducting follow up assessments will be blinded to participant condition in the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Minds Strong Bodies Enhanced (Experimental): The Positive Minds Strong Bodies Enhanced intervention (PMSB-E) consists of 10 sessions focused on mental health (PM) and 36 sessions focused on physical health (SB), along with a group maintenance component.
  Interventions: Behavioral: Positive Minds Strong Bodies Enhanced
- Enhanced Usual Care (Active Comparator): The Enhanced Usual Care condition includes written materials on depression and anxiety and 4 calls to participants over the course of 6 months to assess symptoms and safety.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Positive Minds Strong Bodies Enhanced — The Positive Minds Strong Bodies Enhanced intervention (PMSB-E) was designed to provide a single, integrated program that could address the dual challenges of mental health and disability among minority elders. PMSB-E seeks to improve mood symptoms, identify and correct negative distortions or cognitions, promote behavioral activation through engaging the participant in pleasant activities, and encourage developing supportive relationships. All sessions are tailored to the participant's needs using a collaborative approach.
  Arms: Positive Minds Strong Bodies Enhanced
Behavioral: Enhanced Usual Care — Participants in this arm will receive a booklet about anxiety and depression in Spanish, English, or Mandarin/Cantonese. Research staff will call the participant 4 times over the course of 6 months to administer mental health items, a suicide questionnaire, and a question about medication side effects to mimic the administration schedule in the intervention group.
  Arms: Enhanced Usual Care

SUMMARY:
This study aims to address treatment and service disparities and prevent disability among racial/ethnic and linguistic minority elders. It tests the effectiveness and implementation readiness of the Positive Minds-Strong Bodies Enhanced intervention (PMSB-E), a combined mental and physical health intervention designed to be implemented in low-resource community settings. This renewal grant project includes a streamlined intervention with new components designed to improve and maintain participant outcomes.

DETAILED DESCRIPTION:
The Positive Minds-Strong Bodies Enhanced intervention addresses the dual challenges of mental health and physical disability among minority elders. The core Positive Minds intervention includes 10 sessions offered by Community Health Workers over a maximum of 6 months, designed to identify and correct negative distortions or cognitions, promote behavioral activation and encourage supportive relationships. Strong Bodies is a 36-session physical intervention consisting of a series of exercises conducted while wearing a weighted vest in a group setting over 6 months; both interventions include a group maintenance component to maintain gains. The investigators will evaluate the acceptability, effectiveness and twelve-month sustainability of the Enhanced Positive Minds-Strong Bodies intervention (E-PMSB) offered by Community Health Workers (CHWs) and Exercise Trainers in community-based organizations (CBOs) and community clinics. The intervention is offered in English, Spanish, Mandarin or Cantonese.

ELIGIBILITY:
Inclusion Criteria:

* Latino, Asian, Black, or non-Latino White adults 60+ years of age
* With mild, moderate or severe depressive or anxiety symptoms.
* Participants receiving medications for mental health will have this recorded and used as a covariate.
* Community-dwelling participants who have some mobility limitations but are not home-bound.

Exclusion Criteria:

* Any specialty mental health care (therapy sessions with psychiatrist, psychologist or social worker) in the past 3 months or scheduled in the coming month.
* Evidence that patient lacks capacity to consent or is cognitively impaired
* Current suicidal risk (score of 4 or 5 on Paykel suicide questionnaire), whereby participant will be connected to an emergency services or specialty provider per the study emergency protocol.
* Physically instability, acute or exacerbation of a chronic disease, or a neuro-musculoskeletal impairment
* Severe substance abuse
* Self-reported psychosis or schizophrenia
* Inability to commit to 2 sessions per week

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Acceptability | 6 months at end of treatment
  >/= 70% of participants attending >/= 50% of their intervention sessions, reporting satisfaction with treatment.
Hopkins Symptom Checklist-25 (change) | Baseline and 3, 6, and 12 months after baseline
  Widely used measure of depression and anxiety in clinical monitoring and outcome assessment.
Short Physical Performance Battery (change) | Baseline and 3, 6, and 12 months after baseline
  Assessment of standing balance, timed 4-m walk, and timed test of five chair-rise repetitions, to assess functional limitations. A virtual option will be used while in person assessment is not possible due to COVID-19.
Late-Life Function and Disability Instrument (LLFDI) - functional component (change) | Baseline and 3, 6, and 12 months after baseline
  Self-report instrument designed to measure both functional capacity and components of disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No